CLINICAL TRIAL: NCT04187287
Title: Comparison of Effects of Radial Extracorporeal Shock Wave Therapy and Deep Friction Massage on Individuals With Chronic Lateral Epicondylitis
Brief Title: Comparison of Two Different Treatment Effects on Individuals With Chronic Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Berkiye Kırmızıgil, Director, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/48-01
Record Dates: First submitted 2019-11-29; First posted 2019-12-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Tennis Elbow; Lateral Epicondylitis; Tendinopathy
MeSH Terms: conditions — Tennis Elbow; Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial Extracorporeal Shock Wave Therapy (Active Comparator): Radial Extracorporeal Shock Wave Therapy will be given for 3 weeks, 1 days in a week. Moreover 10-12 minutes cold pack will apply for every session.
  Interventions: Other: Radial Extracorporeal Shock Wave Therapy
- Deep Friction Massage (Active Comparator): Deep Friction Massage treatment will be given for 3 weeks, 3 days in a week. Massage duration will be 10-15 min. for each session. Moreover 10-12 minutes cold pack will apply for every session. Also Mill's manipulation technique will applied once a week during 3 weeks.
  Interventions: Other: Deep Friction Massage

INTERVENTIONS:
Other: Radial Extracorporeal Shock Wave Therapy — Radial Extracorporeal Shock Wave Therapy will given for 3 weeks, 1 days in a week. moreover 10-12 minutes cold pack will apply for every session
  Arms: Radial Extracorporeal Shock Wave Therapy
Other: Deep Friction Massage — Deep Friction Massage will given for 3 weeks, 3 days in a week. Massage duration will be 10-15 min. for each session. Moreover 10-12 minutes cold pack will apply for every session. Also Mill's manipulation technique will applied once a week during 3 weeks.
  Arms: Deep Friction Massage

SUMMARY:
The aim of this study is to compare the effects of Radial Extracorporeal Shockwave Therapy (rESWT) treatment and Deep Friction Massage (DFM) treatment on pain, functionality, grip strength (GS), edema, range of motion (ROM) of the elbow and quality of life in individuals with chronic lateral epicondylitis (CLE).

36 individuals diagnosed with CLE will be randomly divided into two equal groups. rESWT treatment will be applied to Group 1 and DFM treatment to Group 2. Visual analogue scale will be used to assess pain severity, functionality with Patient-Rated Elbow Evaluation Turkish version (PRTEE-T), GS with digital dynamometer, ROM of the elbow joint with goniometer, edema with environmental measurement, and quality of life with Short Form 36 (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with pain on the lateral epicondyle or proximal musculotendinous area of the forearm extensor muscles for at least 3 months,
* Individuals with a positive Thomsen Test ,

  - Individuals who have not received physical therapy for lateral epicondylitis,
* Individuals with a positive Maudsley Test will be included.

Exclusion Criteria:

* Individuals who have received any physical therapy,
* Individuals with reflected pain due to cervical and shoulder pathologies,
* Individuals with elbow osteoarthritis,
* Individuals with previous elbow fractures or elbow joint operations,
* Individuals with a history of systemic inflammatory disease,
* Individuals with osteoporosis,
* Individuals with cardiovascular problems will not be included in the study.

Ages: 20 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Elbow and Forearm Pain | Change from Baseline elbow and forearm pain at 3 weeks
  will assessed using by visual analog scale

SECONDARY OUTCOMES:
Functionality | Change from baseline functionality at 3 weeks
  will assessed using by Patient-Rated Tennis Elbow Evaluation Questionnaire
Grip Strength | Change from baseline grip strength at 3 weeks
  will assessed using by hand grip
Change in the level of elbow and forearm edema | Change from baseline edema at 3 weeks
  Elbow and forearm circumference area will be measured by using a tape measure.
Range of motion of elbow joint | Change from baseline range of motion at 3 weeks
  will evaluated using by goniometer
Change in the level of quality of life | Change from baseline quality of life level at 3 weeks
  will evaluated using by short form 36

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gokalp, Asst. Prof, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus